CLINICAL TRIAL: NCT07039331
Title: The Effects of Short-term Fasting Compared to Free Diet on Ovarian Cancer Patients: A 2-Arms Pilot Randomized Study
Brief Title: Short-term Fasting Compared to Free Diet on Ovarian Cancer Patients
Acronym: DIETA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, MARCHETTI CLAUDIA, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DIETA - ID 3819
Record Dates: First submitted 2025-03-05; First posted 2025-06-26 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a prospective, open-label exploratory randomized clinical trial evaluating the effect of STF on OC patients, receiving NACT with carboplatin and paclitaxel. Potential participants will be screened for eligibility during an appointment at the study center, and eligible candidates will be scheduled for an enrolment appointment. The study physician will perform the candidates' physical examinations. Subjects height and body weight will be measured following a standardized protocol. Body Mass Index (BMI) will be calculated as [weight (kg)] / [height (m)]2. Patient's adverse effects (AE) to the different diets will be recorded on a diary during the entire protocol period.
  Subjects who meet all the inclusion criteria and none of the exclusion criteria will be randomized in a 1:1:1 ratio to one of three arms, as follows:
  * Arm A: Short-Term Fasting
  * Arm B: Free Diet (control arm)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short-Term Fasting (Experimental): Each eligible participant will undergo Short Term Fasting of a total of 60 h during the first three cycles of NACT (36h before and 24h after the end of each cycle of CT).
  Interventions: Dietary Supplement: Short Term Fasting
- Free Diet (Active Comparator): Patients of this group will be invited to follow with their ordinary diet without any change.
  Interventions: Other: Free Diet

INTERVENTIONS:
Dietary Supplement: Short Term Fasting — Short Term Fasting during the first three cycles of NACT (36h before and 24h after the end of each cycle of CT).
  Arms: Short-Term Fasting
Other: Free Diet — Ordinary diet during the first three cycles of NACT without any change.
  Arms: Free Diet

SUMMARY:
The primary endpoint of the study is the reduction of insulin levels between the two groups. Using the Student's t-test, while maintaining the study power at 95% and the significance level at 5%, a sample of 27+27 patients will allow the identification of differences in terms of Cohen's d equal to 1.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effect of STF on OC patients, receiving NACT. The impact on metabolic and endocrine parameters will be investigated, including Insulin level, in order to correlate IGF-1 values and clinical response rate. In particular, the study aims at investigating the reduction in mean insulin levels among different groups (primary endpoint); the effects of the different dietary regimens on metabolic, endocrine, haematologic, inflammatory and tumoral marker response to NACT, the impact of STF on body weight and body composition, ORR, tolerability and toxicity grade experienced by each patient, PFS, QoL and OS will be investigated as secondary clinical outcomes. As translational endpoints, the study will assess the ability of different dietary regimens to modify the immune system; also, the influence of gut microbiota on the chemotherapeutic regimen and on the immune system status in correlation with dietary approach will be explored. Finally, the correlation of intestinal resection during IDS and thereafter the modulation of gut microbiota will be investigated

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 18 years or older;
* Histologically or cytologically documented invasive epithelial OC, primary peritoneal carcinoma, or fallopian tube cancer not suitable for primary cytoreduction, but requiring NACT;
* FIGO Stage III-IV;
* No previous treatment for EOC;
* BMI (Body Mass Index) ≥19 kg/m2;
* ECOG (Eastern Cooperative Oncology Group) performance status 0-2;
* Anticipated life expectancy of >3 months;
* Adequate organ functions:

  * Hematopoietic; Absolute neutrophil count ≥ 1,500/mm^3; Platelet count ≥ 100,000/mm^3; Hemoglobin ≥ 9 g/Dl
  * Hepatic; AST and ALT ≤ 2.5 times upper limit of normal (ULN)* ; Alkaline Phosphatase ≤ 2.5 times ULN* ; Bilirubin ≤ 1.5 times ULN NOTE: * ≤ 3 times ULN if liver metastases are present
  * Renal: Creatinine Clearance ≥ 45 ml/min or Serum Creatinine ≤1.5 x ULN
  * Serum Albumin >2.5 g/dl;
* Patients must be accessible for treatment and follow-up;
* Written informed consent according to the local Ethics Committee requirements
* Patients with child-bearing potential using (or willing to use) effective contraception during treatment and 3 months ahead unless they are postmenopausal (at least 12 months consecutive amenorrhea, in the appropriate age group and without other known or suspected cause), or have been sterilized surgically
* Evidence of not pregnancy status as documented by a negative beta-human chorionic gonadotropin (ß-hCG) test

Exclusion Criteria

* No other invasive malignancy within the past 5 years;
* Diabetes mellitus;
* myocardial infarction, stroke or pulmonary embolism within the last 3 months;
* Electrocardiogram (ECG) demonstrating clinically significant arrhythmias that are not adequately medically managed (Note: subjects with chronic atrial arrhythmia, ie, atrial fibrillation or paroxysmal supraventricular tachycardia [SVT], are eligible)
* Active serious systemic disease, including active bacterial or fungal infection
* Active viral hepatitis or active human immunodeficiency virus (HIV) infection. Asymptomatic positive serology is not exclusionary
* heart failure ≥III NYHA
* Pregnancy or lactating;
* Significant food allergies which would make the subject unable to consume the food provided;
* History of or manifest eating disorder;
* Impaired physical mobility.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 54 (Estimated)
Dates: Start 2021-12-07 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
The effects of short-term fasting and free diet on ovarian cancer | At the end of cycle 3 (each cycle is 21 days)
  The study primary endpoint is the reduction in mean Insulin (µU/ml) levels among different groups.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Marchetti, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- DH Tumori Femminili, Roma, Italy